CLINICAL TRIAL: NCT03739697
Title: Seoul National University Children's Hospital
Brief Title: Effect of Spontaneous Breathing on Atelectasis During Induction of General Anesthesia in Patients in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1810-076-979
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spontaneous breathing (Active Comparator): spontaneous breathing after adminitration of anesthetics
  Interventions: Other: spontaneous breathing
- mechanical ventilation (No Intervention): mechanical ventilation after adminitration of anesthetics and neuromuscula blockade

INTERVENTIONS:
Other: spontaneous breathing — spontaneous breathing during induction of anesthesia in infants
  Arms: spontaneous breathing

SUMMARY:
spontaneous breathing on occurrence of atelectsis in infants

DETAILED DESCRIPTION:
Keeping the spontaneous breathing during the anesthesia for 5 minutes and occurrence of atelectasis

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* heart or lung problems
* prematurity

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
occurrence of atelectasis | 5 minutes after administration of anesthetics
  ateletasis grada (> 2)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji SH, Jang HS, Jang YE, Kim EH, Lee JH, Kim JT, Kim HS. Effect of spontaneous breathing on atelectasis during induction of general anaesthesia in infants: A prospective randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1150-1156. doi: 10.1097/EJA.0000000000001327. PMID 33009186